CLINICAL TRIAL: NCT06407427
Title: Using a Mobile Application for In-Bed Conditioning Exercises for Orthopedic Postoperative Patients
Brief Title: Evaluating the Efficacy of a Mobile Application in Postoperative Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000037597
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Spine Degeneration; Hip Arthritis; Knee Osteoarthritis; Hip Fractures
MeSH Terms: conditions — Osteoarthritis, Knee; Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Care (Experimental): Post-operative usual care where patients will receive standard care plus the use of a tool.
  Interventions: Device: App for in-bed conditioning exercises; Other: Usual care
- Usual Care (Active Comparator): Post-operative usual care where patients will receive standard care alone.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: App for in-bed conditioning exercises — Participants will use an application (app) in facilitating in-bed conditioning exercises for hospitalized patients
  Arms: Enhanced Care
Other: Usual care — All participants will receive usual care in the post-operative setting.

SUMMARY:
This study aims to evaluate the effectiveness of a mobile application in improving postoperative rehabilitation outcomes among patients undergoing orthopedic surgery.

DETAILED DESCRIPTION:
The study aims to assess the effectiveness of a mobile app-based tool in improving conditioning, mobility, and physical therapy performance among patients recovering from orthopedic surgery, particularly hip fracture fixation, spinal fusion, and total knee/hip arthroplasty. The app sets reminders for in-bed conditioning exercises, with difficulty levels adjusted based on patient feedback. The prospective, single-arm pilot study will enroll patients over 65 years old with adequate cognitive status and a mobile phone. Patient performance on the app, satisfaction metrics, and physical therapy outcomes will be evaluated, along with feedback from physical therapists. The study is conducted through the Yale New Haven Health System, with plans to enroll 15 patients initially and subsequently expand to a randomized controlled trial with 50 participants in each arm. The goal is to improve outcomes in this population, characterized by poor mobility, morbidity, and mortality rates, by supplementing inpatient rehabilitation with targeted, app-prompted exercises.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* English reading/speaking
* Are status post low-energy hip fracture, total knee/hip arthroplasty, or single to multilevel spinal fusion without paralysis
* Must be able bodied enough to participate in a mobile app tool for physical therapy
* Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration]

Exclusion Criteria:

* Severe cognitive impairment: Not alert and oriented to person, place, time, and reason for being the hospital; and unable to follow 2 step commands
* Severe physical impairment:

  * Neurologic paralysis
  * Polytraumas with restrictions incompatible with anti-gravity exercises
  * Knee immobilization, bed rest
* Unstable medical conditions:

  * On ventilatory support
  * Utilizing high degrees of oxygen support (continuous BiPAP, high flow nasal cannula, nonrebreather mask, aerosol mask >3L/min)
  * Hemodynamic instability requiring pressor medication support (can include those on pressors for elevated mean arterial pressure goals (MAPs))
  * Neurologically instable with strokes, hemorrhages, increased intracranial pressures
* Open wounds or surgical incisions

  * Tenuous closed wounds requiring immobilization or bending restrictions
  * Open wounds that are either packed/dressed or dressed with a wound vacuum
  * Surgical wounds that are draining fluid or purulence
* Vulnerable populations

  * Incarcerated individuals
* Patients without access to a mobile phone with iOS capability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in patient performance during physical therapy (PT) | Initial (postoperative day 1) and Final PT Visit (at discharge approximately day 3-5 postoperative)
  Patient performance during physical therapy will be assessed using The Activity Measure for Post-Acute Care (AMPAC). The AMPAC score is a comprehensive assessment tool used to evaluate a patient's functional abilities in various domains, including mobility, daily activities, and social interaction. Total score range from 6-24 with higher scores indicating the participant is able to independently perform all activities.

SECONDARY OUTCOMES:
Patient-reported satisfaction metrics | at postoperative day 3-5
  Patients will be surveyed at the end of their intervention using 18 Likert scale (1 to 10), with 10 questions pertaining to their patient care experience, and 8 questions pertaining to their experience using the StrongRx tool. Survey will be piloted to ensure feasibility and ease of completion. Total score range 18-180 with higher scores indicating higher satisfaction.
Length of stay | an average of 3-5 days
  Length of hospital stay serves as a secondary outcome to assess the impact of the intervention on healthcare resource utilization and patient recovery. A shorter length of stay may indicate improved outcomes and efficiency of care delivery, potentially resulting from enhanced rehabilitation efforts facilitated by the tool.
Postoperative VAS scores | immediately postoperative and day of last admission, up to 5 days
  Pain management is a critical aspect of postoperative care, and VAS scores provide a reliable measure of patients' subjective pain levels. Scores will range from 0 (No Pain) to 10 (Worse Pain Possible), with emotion icons to help patients identify which pain level most closely corresponds to their current level. Higher scores indicating more pain.
Patient performance on the app | an average of 3-5 days
  Evaluation of patient performance on the StrongRx app includes tracking points obtained, levels achieved, and exercise sets completed per day. Number of sets completed for each exercise will accrue 1 point for the patient. There will be 3 levels of ease that that will be user directed based on whether the patient is able to easily complete the set. For each level obtained, the points will get a multiplier (1x, 2x, 3x), which corresponds to the multiple of increased repetitions of the exercise. Higher scores indicate more exercises completed.
Patient compliance with prescribed exercises | an average of 3-5 days
  Compliance with prescribed exercises serves to assess the extent to which patients adhere to the recommended rehabilitation regimen. Defined as the number of missed exercises and missed sets.
Physical therapist feedback on app setup assistance, patient interaction, and suggestions for improvement to assess feasibility | up to 120 days
  This data will be gathered as a survey for the physical therapists working on the orthopedics floor at our study site. The survey will include questions regarding the integration of the tool within their workflow, patient interaction, performance during their standardized therapy encounters, and overall recommendation. These will be based on Likert Scale (1 to 10). Total score range 5-50, higher scores indicate more satisfaction. There are also free text questions related to facilitators and barriers.
Adverse Events | Up to 90 Days
  Monitoring adverse events serves as a secondary outcome to evaluate the safety profile of the intervention. Tracking minor events such as hematoma, wound dehiscence, and urinary tract infections, as well as severe events including surgical site infections and pulmonary emboli, provides comprehensive data on potential risks associated with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv S Vasudevan, M.D., Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital Saint Raphael's Campus, New Haven, Connecticut, United States